CLINICAL TRIAL: NCT02645344
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) Combined With Sensory Cueing (SC) on Unilateral Neglect in Subacute Patients With Right Hemispheric Stroke: A Randomized Controlled Study
Brief Title: Effects of Repetitive Transcranial Magnetic Stimulation Combined With Sensory Cueing on Unilateral Neglect in Subacute Patients With Right Hemispheric Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20130720002
Record Dates: First submitted 2015-12-23; First posted 2016-01-01 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Stroke
Keywords: Unilateral neglect; Right hemiplegia
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental): Low frequency rTMS at 1 Hz was applied over P5 of the contralesional hemisphere in addition to conventional rehabilitation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Conventional Rehabilitation
- rTMS combined with sensory cueing (SC) (Experimental): Vibration cueing was emitted using a wristwatch device on the hemiplegic arm combined with low frequency rTMS in addition to conventional rehabilitation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Sensory Cueing (SC); Behavioral: Conventional Rehabilitation
- Conventional rehabilitation (Active Comparator): Physical therapy and occupational therapy
  Interventions: Behavioral: Conventional Rehabilitation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
  Arms: Repetitive Transcranial Magnetic Stimulation (rTMS); rTMS combined with sensory cueing (SC)
Behavioral: Sensory Cueing (SC)
  Arms: rTMS combined with sensory cueing (SC)
Behavioral: Conventional Rehabilitation

SUMMARY:
The objective was to compare the effects of repetitive Transcranial Magnetic Stimulation (rTMS) combined with sensory cueing (SC), rTMS alone, and conventional rehabilitation on reducing unilateral neglect (UN) and improving hemiplegic arm functions and performance of activities of daily living (ADL). Sixty subacute patients with left UN after right-hemispheric stroke were randomly assigned to three groups; rTMS combined with SC, rTMS alone, and conventional rehabilitation. rTMS at 1 Hz was applied over P5 of the contralesional hemisphere while vibration cueing was emitted using a wristwatch device on the hemiplegic arm, five days per week for two weeks. The first two groups received the same dosage of conventional rehabilitation on top of their experimental interventions. Blinded assessments were administered at baseline, 2 weeks postintervention, and four-week follow-up upon completion of training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of right-hemispheric stroke
* Duration since onset of more than one week
* Presenting with unilateral neglect, confirmed by the conventional subtests of the BIT with cutoff scores of 129
* First-ever stroke, or unilateral neglect as the consequence of the last stroke
* Being aged 18 or over
* Mini Mental State Examination score of ≥17
* Giving written consent to participate.

Exclusion Criteria:

* Duration since onset of stroke of more than six months
* Medically unstable
* Epileptic seizures, unconsciousness, or intracranial hypertension
* Serious heart disease
* Gravid
* Severe aphasia so as to have difficulty understanding the therapists' instructions
* Metal implants in vivo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Behavior Inattention Test (BIT) | Change from baseline in 4 weeks (baseline, 2-week and 2-week after training)
Catherine Bergego Scale (CBS) | Change from baseline in 4 weeks (baseline, 2-week and 2-week after training)

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Change from baseline in 4 weeks (baseline, 2-week and 2-week after training)
Action Research Arm Test (ARAT) | Change from baseline in 4 weeks (baseline, 2-week and 2-week after training)
Modified Barthel index (MBI) | Change from baseline in 4 weeks (baseline, 2-week and 2-week after training)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fong KN, Lo PC, Yu YS, Cheuk CK, Tsang TH, Po AS, Chan CC. Effects of sensory cueing on voluntary arm use for patients with chronic stroke: a preliminary study. Arch Phys Med Rehabil. 2011 Jan;92(1):15-23. doi: 10.1016/j.apmr.2010.09.014. PMID 21187201
- [Background] Fong KN, Yang NY, Chan MK, Chan DY, Lau AF, Chan DY, Cheung JT, Cheung HK, Chung RC, Chan CC. Combined effects of sensory cueing and limb activation on unilateral neglect in subacute left hemiplegic stroke patients: a randomized controlled pilot study. Clin Rehabil. 2013 Jul;27(7):628-37. doi: 10.1177/0269215512471959. Epub 2013 Feb 12. PMID 23405025